CLINICAL TRIAL: NCT03018353
Title: Curing HCV in Incarcerated Patients
Acronym: CHIP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: San Francisco Department of Public Health (Other Government)
Collaborators: University of California, San Francisco (Other); San Francisco Study Center (Other); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Lisa Pratt, MD, Medical Director, Jail Health Services, San Francisco Department of Public Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-337-1941
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Jail; Patient Navigation; Incarcerated Population; HCV; Sofosbuvir/Velpatasvir; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Navigation services with sof/vel therapy (Other): This a single group demonstration project in which, patients are treated with the FDA-approved drug, Sofosbuvir/Velpatasvir (Epclusa). If a patients is released during their treatment regimen, they will receive patient navigation services to continue their care and treatment in the community.
  Interventions: Drug: Patients receiving Sof/Vel (Epclusa) and Navigation services

INTERVENTIONS:
Drug: Patients receiving Sof/Vel (Epclusa) and Navigation services — Implementing HCV treatment in the jails using FDA-approved medications and continuing there treatment in the community if they are released during their treatment regimen.

SUMMARY:
Curing HCV in Incarcerated Patients (CHIP) is a 1-year demonstration project that will assess the feasibility of a HCV treatment program in the San Francisco City & County Jail. The Jail Health Services will treat 100 patients using the FDA approved combination treatment, sofosbuvir/velpatasvir, Epclusa® and will continue their treatment during incarceration and after their release (if applicable).

DETAILED DESCRIPTION:
Curing HCV in Incarcerated Patients (CHIP) is a 1-year demonstration project that will be conducted in the San Francisco County Jails. Jail settings can provide an optimal opportunity to screen for HCV, initiate curative treatment, and link patients to community HCV providers to complete their treatment. This demonstration project will be funded by the Gilead's Investigator Sponsored Research. The purpose is to assess the feasibility of treating inmates with the FDA approved combination oral treatment, sofosbuvir/velpatasvir, Epclusa®. The San Francisco Department of Public Health's Jail Health Services will treat 100 patients. Intensive patient navigators will be an essential component for treatment to ensure medication adherence and achieve SVR for those who are discharged from jail prior to HCV treatment completion. Navigators will provide short-term case management services by linking patients to medical and social support services. This demonstration project will be facilitated by the Jail Health Services' HIV & Integrated Services (formerly Forensic AIDS Project).

ELIGIBILITY:
Inclusion Criteria:

* a detectable HCV viral load
* no medical contraindications to treatment, including limited life expectancy of less than 12-months due to non-liver related comorbid conditions or renal failure with creatinine clearance of < 30 mL/min.
* Must start HCV treatment while detained
* HIV positive or negative status
* HBV positive or negative status
* treatment-naïve or experienced
* with or without cirrhosis

Exclusion Criteria:

* a limited life expectancy of less than 12-months due to non-liver related comorbid conditions
* current or history of decompensated cirrhosis, defined as presence of ascites, hepatic encephalopathy, or variceal bleeding within the past 6 months.
* severe renal impairment defined as creatinine clearance of < 30 mL/min or end stage renal disease (ESRD) on hemodialysis
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-03-05 (Actual); Primary Completion 2018-03-04 (Estimated); Study Completion 2018-06-04 (Estimated)

PRIMARY OUTCOMES:
SVR12 of 70% or greater | 12 months
  The primary objective is to implement a feasible HCV treatment program in an urban jail setting, City & County of San Francisco, over a 12 month period, with demonstration of a SVR12 of 70% or greater among inmates who initiates HCV treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Jail Health Services, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other outside researchers who are not participating in this pilot demonstration project.